CLINICAL TRIAL: NCT00961532
Title: Improving Platelet Activity for Cerebral Hemorrhage Treatment - DDAVP Proof of Concept
Acronym: IMPACT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Northwestern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Andrew Naidech, Associate Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU8168
Record Dates: First submitted 2009-08-17; First posted 2009-08-19 (Estimated); Results first posted 2014-08-28 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-07

CONDITIONS: Intracerebral Hemorrhage
Keywords: intracerebral hemorrhage; platelets
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Deamino Arginine Vasopressin

ARMS (1):
- DDAVP (Experimental): DDAVP 0.4 mcg/kg intravenously in 250 mL NS over 30 minutes
  Interventions: Drug: DDAVP injection (desmopressin acetate)

INTERVENTIONS:
Drug: DDAVP injection (desmopressin acetate) — 0.4 mcg/kg in 250 mL NS intravenously once over 30 minutes

SUMMARY:
The investigators intend to show that DDAVP improves platelet activity from baseline to 60 minutes after treatment start.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous intracerebral hemorrhage as documented by head CT scan
* Documented regular aspirin use or VerifyNow-ASA result of ≤ 550 aspirin reaction units (ARU), indicating anti-platelet medication

Exclusion Criteria:

* International normalized ratio (INR) of ≥ 1.7 from coagulopathy or warfarin use
* History of von Willebrand disease
* Pregnancy
* Known hypersensitivity to DDAVP or desmopressin
* Active cardiovascular disease or unstable angina
* Hyponatremia or history of hyponatremia
* Current or historical deep venous thrombosis or pulmonary embolism

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Naidech, MD MSPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Result] Naidech AM, Maas MB, Levasseur-Franklin KE, Liotta EM, Guth JC, Berman M, Rosenow JM, Lindholm PF, Bendok BR, Prabhakaran S, Bernstein RA, Kwaan HC. Desmopressin improves platelet activity in acute intracerebral hemorrhage. Stroke. 2014 Aug;45(8):2451-3. doi: 10.1161/STROKEAHA.114.006061. Epub 2014 Jul 8. PMID 25005444

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DDAVP
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | DDAVP
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Platelet Activity, Measured in Seconds on PFA-EPI Assay, From Pre to Post-treatment
Description: The Platelet Function Analyzer (PFA) is a commercially available point-of-care assay that measures the time to closure of an aperature. Longer time to closure indicates less platelet activity. EPI denotes epinephrine (as opposed to adenosine diphosphate) as the stimulant to platelet aggregation. In our laboratory, a time to closure of at least 172 seconds in consistent with an aspirin effect.
Time Frame: 60 minutes after treatment start
Measure: Mean (Standard Error); unit: seconds
Arm/Group | DDAVP
Number analyzed (Participants) | 14
seconds | 68 (24.1)
Statistical Analysis 1: Comparison: DDAVP; We tested the hypothesis that there would be a change from baseline to 60 minutes after the start of the desmopressin (DDAVP) infusion; Test type: Superiority or Other; p = 0.014, t-test, 2 sided

2. Secondary Outcome: Adverse Events : New Fever >=100.4F, Respiratory Distress or Pulmonary Edema on Chest Radiography, Rash, Hypotension (Systolic BP < 100 mm Hg or New Vasopressor Use or Increase in Vasopressor Dose by >25%)
Description: We prospectively defined acute adverse events as: new fever >=100.4F, respiratory distress or pulmonary edema on chest radiography, rash, hypotension (systolic BP < 100 mm Hg or new vasopressor use or increase in vasopressor dose by >25%). The two patients reported were the only two that sustained any of the prospectively defined adverse events.
Time Frame: within 6 hours of study treatment
Measure: Number; unit: participants
Arm/Group | DDAVP
Number analyzed (Participants) | 14
participants | 2

ADVERSE EVENTS:
Arm/Group | DDAVP
Serious Adverse Events (participants affected / at risk) | 2/14
Other Adverse Events (participants affected / at risk) | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DDAVP (N=14)
Hypotension (Cardiac disorders) | 1
Fever (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No